CLINICAL TRIAL: NCT02152995
Title: A Phase 2 Study of Trametinib in Combination With Radioiodine (RAI) for RAS Mutant or RAS/RAF Wild-Type, RAI-Refractory Recurrent and/or Metastatic Thyroid Cancers
Brief Title: Trametinib in Increasing Tumoral Iodine Incorporation in Patients With Recurrent or Metastatic Thyroid Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-01106; NCI-2014-01106 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-157; 9446 (Other: Memorial Sloan Kettering Cancer Center); 9446 (Other: CTEP); P30CA008748 (NIH); P50CA172012 (NIH); R01CA184724 (NIH)
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Results first posted 2022-12-28 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Thyroid Gland Carcinoma; Poorly Differentiated Thyroid Gland Carcinoma; Recurrent Thyroid Gland Carcinoma; Refractory Thyroid Gland Carcinoma; Stage IV Thyroid Gland Follicular Carcinoma AJCC v7; Stage IV Thyroid Gland Papillary Carcinoma AJCC v7; Stage IVA Thyroid Gland Follicular Carcinoma AJCC v7; Stage IVA Thyroid Gland Papillary Carcinoma AJCC v7; Stage IVB Thyroid Gland Follicular Carcinoma AJCC v7; Stage IVB Thyroid Gland Papillary Carcinoma AJCC v7; Stage IVC Thyroid Gland Follicular Carcinoma AJCC v7; Stage IVC Thyroid Gland Papillary Carcinoma AJCC v7
MeSH Terms: conditions — Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary | interventions — Iodine-124; Iodine-131; Magnetic Resonance Spectroscopy; trametinib; omipalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort A (iodine I-124 PET/CT, trametinib, iodine I-131) (Experimental): Patients with RAS gene mutations undergo iodine I-124 PET/CT on day 5 of week 1. Beginning day 6, patients receive trametinib PO daily for 4 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo second iodine I-124 PET/CT on week 5. If I-124 PET/CT shows enough iodine absorption, patients may receive iodine I-131 PO and continue receiving trametinib for another 2 days. If I-124 shows that the thyroid is not absorbing iodine, patients have the option to be assigned to Cohort C.
  Interventions: Procedure: Computed Tomography; Other: Iodine I 124; Radiation: Iodine I-131; Other: Laboratory Biomarker Analysis; Other: Pharmacodynamic Study; Procedure: Positron Emission Tomography; Drug: Trametinib
- Cohort B (iodine I-124 PET/CT, trametinib, iodine I-131) (Experimental): Patients without BRAF/RAS gene mutations undergo iodine I-124 PET/CT on day 5 of week 1. Beginning day 6, patients receive trametinib PO daily for 4 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo second iodine I-124 PET/CT on week 5. If I-124 PET/CT shows enough iodine absorption, patients may receive iodine I-131 PO and continue receiving trametinib for another 2 days. If I-124 shows that the thyroid is not absorbing iodine, patients have the option to be assigned to Cohort C.
  Interventions: Procedure: Computed Tomography; Other: Iodine I 124; Radiation: Iodine I-131; Other: Laboratory Biomarker Analysis; Other: Pharmacodynamic Study; Procedure: Positron Emission Tomography; Drug: Trametinib
- Cohort C (trametinib) (Experimental): Patients may continue trametinib at the doctor's discretion and do not receive iodine I-131.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacodynamic Study; Drug: Trametinib

INTERVENTIONS:
Procedure: Computed Tomography — Undergo iodine I-124 PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
  Arms: Cohort A (iodine I-124 PET/CT, trametinib, iodine I-131); Cohort B (iodine I-124 PET/CT, trametinib, iodine I-131)
Other: Iodine I 124 — Undergo iodine I-124 PET/CT
  Other Names: I-124; Iodine 124; Iodine I-124
  Arms: Cohort A (iodine I-124 PET/CT, trametinib, iodine I-131); Cohort B (iodine I-124 PET/CT, trametinib, iodine I-131)
Radiation: Iodine I-131 — Given PO
  Other Names: 131-Iodine; Bound Iodide I-131; I 131; I-131; Iodide I-131; Iodide, I-131; Iodine 131; Iodine-131; Iodotope; Iodotrope
  Arms: Cohort A (iodine I-124 PET/CT, trametinib, iodine I-131); Cohort B (iodine I-124 PET/CT, trametinib, iodine I-131)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacodynamic Study — Correlative studies
  Other Names: PHARMACODYNAMIC; Pharmacodynamic (PD) study
Procedure: Positron Emission Tomography — Undergo iodine I-124 PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
  Arms: Cohort A (iodine I-124 PET/CT, trametinib, iodine I-131); Cohort B (iodine I-124 PET/CT, trametinib, iodine I-131)
Drug: Trametinib — Given PO
  Other Names: GSK 1120212; GSK 212; GSK-1120212; GSK-212; GSK1120212; GSK212; JTP 74057; JTP-74057; JTP74057; MEK Inhibitor GSK1120212

SUMMARY:
This phase II trial studies how well trametinib works in increasing tumoral iodine incorporation in patients with thyroid cancer that has come back or spread to another place in the body. Trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and may help make treatment with iodine I-131 more effective.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect of trametinib on enhancing radioiodine (RAI) activity by determining the proportion of patients alive at 6 months without disease progression by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST version [v]1.1) criteria following treatment with RAI in co-administration with trametinib. (Cohort A) II. To evaluate the effect of trametinib on enhancing RAI activity by determining the objective response rate (ORR) at 6 months following treatment with radioiodine (RAI) in co-administration with trametinib. (Cohort A) III. To determine the proportion of patients following trametinib therapy with increased tumoral iodine incorporation as quantified by iodine iodine-124 (I-124) positron emission tomography (PET)/computed tomography (CT) lesional dosimetry. (Cohort B)

SECONDARY OBJECTIVES:

I. To determine the proportion of patients following trametinib therapy with increased tumoral iodine incorporation as quantified with I-124 PET/CT lesional dosimetry. (Cohort A) II. To evaluate the safety/tolerability of trametinib with or without RAI. (Cohort A) III. To evaluate changes in thyroglobulin levels in patients treated with RAI. (Cohort A) IV. To explore potential correlations between genomic alterations present in the tumor and/or tumoral pharmacodynamic changes induced by trametinib to clinical outcomes. (Exploratory) (Cohort A) V. To evaluate the effect of trametinib on enhancing RAI activity by determining the ORR at 6 months following treatment with RAI in co-administration with trametinib. (Cohort B) VI. To evaluate the effect of trametinib on enhancing RAI activity by determining the proportion of patients alive at 6 months without disease progression by RECIST v 1.1 criteria following treatment with RAI in co-administration with trametinib. (Cohort B) VII. To evaluate the safety/tolerability of trametinib with or without RAI. (Cohort B) VIII. To evaluate changes in thyroglobulin levels in patients treated with RAI. (Cohort B) IX. To explore potential correlations between genomic alterations present in the tumor and/or tumoral pharmacodynamic changes induced by trametinib to clinical outcomes. (Exploratory) (Cohort B) X. Preliminary evaluation of best objective response (BOR) rate for patients treated with trametinib alone. (Exploratory) (Cohort C) XI. Preliminary evaluation of the proportion of patients following treatment with trametinib alive at 6 months without disease progression by RECIST v 1.1 criteria. (exploratory) (Cohort C) XII. To evaluate the safety/tolerability of trametinib. (Cohort C) XIII. To evaluate changes in thyroglobulin levels in patients treated with trametinib. (Cohort C) XIV. To explore potential correlations between genomic alterations present in the tumor and/or tumoral pharmacodynamic changes induced by trametinib to clinical outcomes. (Exploratory) (Cohort C) XV. To explore the impact of continued trametinib upon RAI avidity and efficacy. (Exploratory) (Cohort C)

OUTLINE: Patients with RAS gene mutations are assigned to Cohort A, while patients without BRAF/RAS gene mutations are assigned to Cohort B.

COHORT A: Patients undergo iodine I-124 PET/CT on day 5 of week 1. Beginning day 6, patients receive trametinib orally (PO) daily for 4 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo second iodine I-124 PET/CT on week 5. If I-124 PET/CT shows enough iodine absorption, patients may receive iodine I-131 PO and continue receiving trametinib for another 2 days. If I-124 shows that the thyroid is not absorbing iodine, patients have the option to be assigned to Cohort C.

COHORT B: Patients undergo iodine I-124 PET/CT on day 5 of week 1. Beginning day 6, patients receive trametinib PO daily for 4 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo second iodine I-124 PET/CT on week 5. If I-124 PET/CT shows enough iodine absorption, patients may receive iodine I-131 PO and continue receiving trametinib for another 2 days. If I-124 shows that the thyroid is not absorbing iodine, patients have the option to be assigned to Cohort C.

COHORT C: Patients may continue trametinib at the doctor's discretion and do not receive iodine I-131.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed thyroid carcinoma of follicular origin (including papillary, follicular, or poorly differentiated subtypes and their respective variants); confirmation of thyroid carcinoma will be done at Memorial Sloan-Kettering (MSK)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan, magnetic resonance imaging (MRI), or calipers by clinical exam; tumors in previously irradiated fields may be considered measurable if there is evidence of tumor progression after radiation treatment
* RAI-refractory disease on structural imaging, defined as any one of the following:

  * A metastatic lesion that is not radioiodine-avid on a diagnostic radioiodine scan performed prior to enrollment in the current study, or
  * A radioiodine-avid metastatic lesion which remained stable in size or progressed despite radioiodine treatment 6 months or more prior to entry in the study; there are no size limitations for the index lesion used to satisfy this entry criterion
  * The presence of at least one fluorodeoxyglucose (FDG) avid lesion
* No recent treatment for thyroid cancer as defined as:

  * No prior RAI therapy is allowed < 6 months prior to initiation of therapy on this protocol; a diagnostic study using < 10 millicurie (mCi) of RAI is not considered RAI therapy
  * No external beam radiation therapy < 4 weeks prior to initiation of therapy on this protocol; (previous treatment with radiation for any indication is allowed if the investigator judges that the previous radiation does not significantly compromise patient safety on this protocol)
  * No chemotherapy or targeted therapy (e.g., tyrosine kinase inhibitor) is allowed < 4 weeks prior to the initiation of therapy on this protocol
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Able to swallow and retain orally-administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* All prior treatment-related toxicities must be Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v 4.0) grade =< 1 (except alopecia); grade 2 prior treatment related toxicities may be allowed after discussion with the principal investigator
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Hemoglobin >= 9 g/dL
* Platelets >= 100 x 10^9/L
* Albumin >= 2.5 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional ULN
* Creatinine =< 1.5 mg/dL OR calculated creatinine clearance (Cockcroft-Gault formula) >= 50 mL/min OR 24-hour urine creatinine clearance >= 50 mL/min
* Prothrombin time (PT) or international normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 x institutional ULN
* Left ventricular ejection fraction >= institutional lower limit of normal (LLN) by echocardiogram (ECHO) or multi gated acquisition scan (MUGA)
* The effects of trametinib on the developing human fetus are unknown; since MEK inhibitors and RAI may be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study, and 4 months after study completion; women of child-bearing potential must have a negative pregnancy test within 2 weeks prior study registration; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform the treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of trametinib administration
* Ability to understand and the willingness to sign a written informed consent document
* Patients must agree to undergo two separate biopsies of a malignant lesion; biopsies do not need to be done if one of the following apply:

  * If either the site investigator or person performing the biopsy judges that no tumor is accessible for biopsy or that biopsy poses too great of a risk to the patient (if the only tumor accessible for biopsy is also the only lesion that can be used for RECIST v1.1 response evaluation, then the patient may be exempt from biopsy after discussion with the MSK principal investigator)
  * The goal will be to have a minimum of 6 patients from Cohort A and 3 patients from Cohort B attempt to have one or both of these research biopsies done (for a total of 9 patients total); accrual may be limited only to subjects for whom tumor is accessible for biopsy and attempt at biopsy is considered safe if continued enrollment of those who are not candidates for biopsy make it impossible to reach the accrual goals for research biopsies described above (e.g., if 19 [of 25] patients are accrued to Cohort A without any biopsies having been obtained within the cohort, then all further subjects who are registered to that cohort must qualify for attempted research biopsy in order to be enrolled into the study [i.e., subjects who would have been excluded from having biopsies done due to the above reasons would be excluded from participating in the study; these conditions also apply to Cohort B])
* Availability of archival tumor tissue from the thyroid cancer primary or metastasis (a tissue block or a minimum of 30 unstained slides would be required; patients with less archival tissue available may still be eligible for the study after discussion with the MSK principal investigator)
* COHORT A: Confirmation in a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory that one of the patient's thyroid tumors (primary tumor, recurrent tumor, or metastasis) has an neuroblastoma RAS viral (v-ras) oncogene homolog (NRAS) or Kirsten rat sarcoma viral oncogene homolog (KRAS) or Harvey rat sarcoma viral oncogene homolog (HRAS) mutation at G12, G13, or Q61; this group of patients will also be referred to as "RAS MUT"
* COHORT A: Patients must have progressive disease, defined as the presence of new or growing lesion(s) on radiologic imaging within 14 months of study enrollment and/or new/worsening disease related symptoms within 14 months of study enrollment; (progression according to RECIST v 1.1 criteria is not required)
* COHORT B: Confirmation in a CLIA certified laboratory that one of the patient's thyroid tumors (primary tumor, recurrent tumor, or metastasis) does not have any of the following mutations:

  * Mutation at V600 of the v-raf murine sarcoma viral oncogene homolog B (BRAF) gene
  * Mutation in NRAS or KRAS or HRAS at G12, G13, or Q61
  * These patients will be designated "BRAF/RAS wild type (WT)"

Exclusion Criteria:

* History of another malignancy; exception: patients who have been disease-free for 3 years, patients with a history of completely resected non-melanoma skin cancer, and/or patients with indolent secondary malignancies, are eligible; MSK can consult the Cancer Therapy Evaluation Program (CTEP) Medical Monitor if unsure whether second malignancies meet the requirements specified above
* History of interstitial lung disease or pneumonitis
* Use of other investigational drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of trametinib and during the study
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trametinib, or excipients or to dimethyl sulfoxide (DMSO) or to thyrotropin alpha (Thyrogen)
* Current use of a prohibited medication; the following medications or non-drug therapies are prohibited:

  * Other anti-cancer therapy while on study; (note: megestrol [Megace] if used as an appetite stimulant is allowed; thyroid-stimulating hormone [TSH] suppressive therapy is also allowed; palliative radiation therapy to non-target lesions is also allowed)
  * Concurrent treatment with bisphosphonates is permitted; prophylactic use of bisphosphonates in patients without bone disease is not permitted, except for the treatment of osteoporosis
  * Because the composition, pharmacokinetics (PK), and metabolism of many herbal supplements are unknown, the concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, St. John's wort, kava, ephedra [ma huang], gingko biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, or ginseng)
* Patients with the following ophthalmological findings/conditions:

  * Intraocular pressure > 21 mmHg, or uncontrolled glaucoma (irrespective of intraocular pressure)
  * Current or past history of central serious retinopathy or retinal vein occlusion
* History or evidence of cardiovascular risk including any of the following:

  * Left ventricular ejection fraction (LVEF) < LLN
  * A QT interval corrected for heart rate using the Bazett's formula (QTcB) >= 480 msec
  * History or evidence of current clinically significant uncontrolled arrhythmias (exception: patients with controlled atrial fibrillation for > 30 days prior to randomization are eligible)
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization
  * History or evidence of current >= class II congestive heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Treatment-refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy
  * Patients with intra-cardiac defibrillators
  * Known cardiac metastases
* Known human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection (with the exception of chronic or cleared HBV and HCV infection, which will be allowed); patients with human immunodeficiency virus (HIV) are not eligible if on anti-retroviral medications
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Animal reproductive studies have not been conducted with trametinib; therefore, the study drug must not be administered to pregnant women or nursing mothers; these potential risks may also apply to RAI and Thyrogen
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with trametinib; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy
* Patients unable to follow a low iodine diet or requiring medication with high content in iodide (amiodarone)
* Patients who received iodinated intravenous contrast as part of a radiographic procedure within 3 months of study registration; those that have had iodinated intravenous contrast within this time frame may still be eligible if a urinary iodine analysis reveals that the excess iodine has been cleared after the last intravenous contrast administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-08-14 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2026-01-25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alan L Ho, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A (Iodine I-124 PET/CT, Trametinib, Iodine I-131) | Cohort B (Iodine I-124 PET/CT, Trametinib, Iodine I-131)
Started | 25 | 9
Participants Who Continued Treatment With Trametinib Only | 5 | 2
Completed | 24 | 9
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Iodine I-124 PET/CT, Trametinib, Iodine I-131) | Cohort B (Iodine I-124 PET/CT, Trametinib, Iodine I-131) | Total
Number analyzed (Participants) | 25 | 9 | 34
Age, Continuous [Mean (Full Range); unit: years] | 53.2 [27 to 73] | 53.4 [31 to 69] | 53.3 [27 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14
  Male | 15 | 5 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 24 | 9 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 19 | 8 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 9 | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Progression Free at 6 Months Following Treatment With Trametinib and I-124 (Cohort A)
Description: Cohort A only. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: At 6 months
Measure: Number; unit: % of pts progression free at 6 months
Arm/Group | Cohort A (Iodine I-124 PET/CT, Trametinib, Iodine I-131)
Number analyzed (Participants) | 25
% of pts progression free at 6 months | 44

2. Primary Outcome: Progression Free Survival (Cohort A)
Description: An exact binomial stage design will be used to discriminate between true 6-month progression/death rates of 20% vs 50%, and between true ORR rates at 6 months of 5% and 25%. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Iodine I-124 PET/CT, Trametinib, Iodine I-131)
Number analyzed (Participants) | 25
Participants
  Pts progression-free at 6 months | 11
  Pts who were not progression-free at 6 months | 14

3. Primary Outcome: Percentage With Objective Response (Complete Response or Partial Response) (Cohort A)
Description: Will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. An exact binomial stage design will be used to discriminate between true 6-month ORR rates at 6 months of 5% and 25%. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: At 6 months
Measure: Number; unit: % of pts with confirmed partial response
Arm/Group | Cohort A (Iodine I-124 PET/CT, Trametinib, Iodine I-131)
Number analyzed (Participants) | 25
% of pts with confirmed partial response | 32

4. Primary Outcome: Iodine Incorporation in Thyroid Cancer Metastases to a Predicted Lesional Absorbed Radiation Dose Equal to or Exceeding 2,000 cGy With the Administration of =< 300 mCi Radioiodine (RAI) (Cohort B)
Description: "Adequate increase" is defined as increasing iodine incorporation in thyroid cancer metastases to a predicted lesional absorbed radiation dose equal to or exceeding 2,000 cGy with the administration of < 300 mCi RAI. Iodine incorporation is quantified with PET/CT lesional dosimetry.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B (Iodine I-124 PET/CT, Trametinib, Iodine I-131)
Number analyzed (Participants) | 9
Participants
  Pts who met the lesional dosimetry threshold for I-131 therapy | 4
  Pts who did not meet the lesional dosimetry threshold for I-131 therapy | 5

5. Secondary Outcome: Adequate Increase in Iodine Corporation (Cohort A)
Description: Will be determined by treatment with trametinib in thyroid cancer metastases to a predicted lesional absorbed radiation dose equal to or exceeding 2,000 cGy with the administration of =< 300 mCi radioiodine (RAI). Proportion of patients with an adequate increase will be reported, along with the corresponding exact 95% confidence interval.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Iodine I-124 PET/CT, Trametinib, Iodine I-131)
Number analyzed (Participants) | 25
Participants
  Pts who met the lesional dosimetry threshold for I-131 therapy | 15
  Pts who did not meet the lesional dosimetry threshold for I-131 therapy | 10

6. Secondary Outcome: Changes in Thyroglobulin
Description: Wilcoxon signed rank test will be performed for paired samples to compare the thyroglobulin level before and after RAI treatment in the subset of patients treated with RAI.
Time Frame: Baseline to up to 6 months
Population: Data were not collected
Arm/Group | Cohort A (Iodine I-124 PET/CT, Trametinib, Iodine I-131) | Cohort B (Iodine I-124 PET/CT, Trametinib, Iodine I-131)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Toxicity (Cohort A)
Description: Will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Toxicities will be individually reported and summarized.
Time Frame: Up to 30 days after completion of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Iodine I-124 PET/CT, Trametinib, Iodine I-131)
Number analyzed (Participants) | 25
Participants | 25

8. Secondary Outcome: Percentage With an Objective Response (Complete Response or Partial Response) (Cohort B)
Description: Will be assessed by RECIST v1 1.1 criteria. An exact binomial stage design will be used to discriminate between true 6-month ORR rates at 6 months of 5% and 25%.
Time Frame: At 6 months
Measure: Number; unit: % of pts with confirmed partial response
Arm/Group | Cohort B (Iodine I-124 PET/CT, Trametinib, Iodine I-131)
Number analyzed (Participants) | 9
% of pts with confirmed partial response | 11

9. Secondary Outcome: Percentage of Patients Alive Without Disease Progression (Cohort B)
Description: Assessed per RECIST v1.1. Will be estimated using 95% confidence intervals.
Time Frame: At 6 months
Measure: Number; unit: % of pts progression free at 6 months
Arm/Group | Cohort B (Iodine I-124 PET/CT, Trametinib, Iodine I-131)
Number analyzed (Participants) | 9
% of pts progression free at 6 months | 44

10. Secondary Outcome: Change in Thyroglobulin (Cohort B)
Description: Will determine whether treatment with trametinib and RAI results in decreasing thyroglobulin. Will perform a Wilcoxon signed rank test for paired samples to compare the thyroglobulin level before and after RAI treatment in the subset of patients treated with RAI.
Time Frame: Baseline up to 6 months
Population: Data were not collected
Arm/Group | Cohort B (Iodine I-124 PET/CT, Trametinib, Iodine I-131)
Number analyzed (Participants) | 0

11. Secondary Outcome: Number of Participants With Toxicity (Cohort B)
Description: Will be assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.0. Toxicities will be individually reported and summarized. Beginning April 1, 2018, CTCAE v5.0 will be utilized for adverse event (AE) reporting.
Time Frame: Up to 30 days after completion of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B (Iodine I-124 PET/CT, Trametinib, Iodine I-131)
Number analyzed (Participants) | 9
Participants | 9

12. Other Pre Specified Outcome: Expression and Phosphorylation of MAPK Signaling Pathway Proteins
Description: Analyses will be descriptive.
Time Frame: Up to 6 months
Population: Data were not collected
Arm/Group | Cohort A (Iodine I-124 PET/CT, Trametinib, Iodine I-131) | Cohort B (Iodine I-124 PET/CT, Trametinib, Iodine I-131)
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Expression and Phosphorylation of Negative Feedback Loops Connected to the MAPK Pathway (Such as Human Epidermal Growth Factor 3)
Description: Analyses will be descriptive.
Time Frame: Up to 6 months
Population: Data were not collected
Arm/Group | Cohort A (Iodine I-124 PET/CT, Trametinib, Iodine I-131) | Cohort B (Iodine I-124 PET/CT, Trametinib, Iodine I-131)
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Quantitative Levels of Messenger Ribonucleic Acid Transcripts for MAPK Regulated and Thyroid-specific Gene Products
Description: Analyses will be descriptive.
Time Frame: Up to 6 months
Population: Data were not collected
Arm/Group | Cohort A (Iodine I-124 PET/CT, Trametinib, Iodine I-131) | Cohort B (Iodine I-124 PET/CT, Trametinib, Iodine I-131)
Number analyzed (Participants) | 0 | 0

15. Other Pre Specified Outcome: Presence of Other Genetic Alterations
Description: Analyses will be descriptive.
Time Frame: Up to 6 months
Population: Data were not collected
Arm/Group | Cohort A (Iodine I-124 PET/CT, Trametinib, Iodine I-131) | Cohort B (Iodine I-124 PET/CT, Trametinib, Iodine I-131)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Cohort A (Iodine I-124 PET/CT, Trametinib, Iodine I-131) | Cohort B (Iodine I-124 PET/CT, Trametinib, Iodine I-131)
All-Cause Mortality (participants affected / at risk) | 6/25 | 1/9
Serious Adverse Events (participants affected / at risk) | 6/25 | 1/9
Other Adverse Events (participants affected / at risk) | 25/25 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (Iodine I-124 PET/CT, Trametinib, Iodine I-131) (N=25) | Cohort B (Iodine I-124 PET/CT, Trametinib, Iodine I-131) (N=9)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Ejection Fraction Decrease (Cardiac disorders) | 0 | 0
Death NOS (General disorders) | 6 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (Iodine I-124 PET/CT, Trametinib, Iodine I-131) (N=25) | Cohort B (Iodine I-124 PET/CT, Trametinib, Iodine I-131) (N=9)
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Alanine aminotransferase increased (Investigations) | 7 | 0
Alkaline phosphatase increased (Investigations) | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0
Anemia (Blood and lymphatic system disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 15 | 2
Blurred vision (Eye disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 7 | 5
Dry mouth (Gastrointestinal disorders) | 6 | 1
Dysgeusia (Nervous system disorders) | 4 | 0
Edema limbs (General disorders) | 5 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Fatigue (General disorders) | 14 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Gen disorders & admin site conditions Other, spec (General disorders) | 1 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypertension (Vascular disorders) | 8 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 10 | 3
Oral pain (Gastrointestinal disorders) | 1 | 1
Pain (General disorders) | 1 | 1
Paresthesia (Nervous system disorders) | 0 | 2
Platelet count decreased (Investigations) | 8 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 12 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 | 3
Vomiting (Gastrointestinal disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/95/NCT02152995/Prot_SAP_000.pdf